CLINICAL TRIAL: NCT01270295
Title: Soluble Forms and Ligands of the Receptor for Advanced Glycation End Products (RAGE) in the Pulmonary Edema Fluid and Plasma From ICU Patients With ALI/ARDS : an Observational Prospective Study.
Brief Title: Soluble Forms and Ligands of RAGE in ALI/ARDS (SoLiRAGE).
Acronym: SoLiRAGE
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0086
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome; Mechanical Ventilation
Keywords: Receptor for advanced glycation end products (RAGE); Soluble RAGE (sRAGE); Endogenous secretory RAGE (esRAGE); High-mobility group box-1 protein (HMGB-1); Extracellular newly-identified RAGE-binding protein (EN-RAGE or S100A12); Advanced glycation endproducts (AGEs); Pentosidine; N--carboxymethyllysine; Acute lung injury (ALI); Acute respiratory distress syndrome (ARDS); Alveolar epithelium; Mechanical ventilation; Intensive Care Unit (ICU)
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
RAGE, the receptor for advanced glycation end products, is a novel marker of alveolar epithelial type I cell injury. Soluble RAGE (sRAGE) is elevated in the plasma and in the pulmonary edema fluid from patients with ALI/ARDS, but one should acknowledge that the RAGE/NF-B axis is also involved in the pathophysiology of various other conditions. Few data are available about the levels of soluble forms and ligands of RAGE in the setting of ALI/ARDS. The purpose of this observational prospective study is to describe soluble forms (sRAGE, esRAGE) and ligands of RAGE (HMGB-1, S100A12, AGEs) levels in ICU patients with ALI/ARDS.

DETAILED DESCRIPTION:
BACKGROUND:

The receptor for advanced glycation end products (RAGE) is now identified as a marker of alveolar type I cell injury. RAGE is a member of the immunoglobulin superfamily that acts as a multiligand receptor and is involved in propagating inflammatory responses. While the precise function of RAGE remains unclear, the elevated levels of RAGE, and its soluble isoform sRAGE, correlate with severity of ALI/ARDS in human and animal studies, and RAGE levels could reflect impaired alveolar fluid clearance. Frequently, the biology of RAGE coincides with settings in which ligands of the receptor accumulate, especially in a proinflammatory environment. More work is needed for us to understand the mechanisms by which RAGE is regulated during ALI/ARDS, especially with regard to the expression of its soluble forms and the involvement of its potential ligands.

DESIGN NARRATIVE:

This observational prospective clinical study will describe and compare soluble forms (sRAGE, esRAGE) and ligands of RAGE (HMGB-1, S100A12, AGEs) levels in the alveolar edema fluid and in the plasma from ICU patients enrolled within the first 24 hours after onset of ALI/ARDS, and from patients under mechanical ventilation (control group).

Edema fluid and plasma samples will be collected simultaneously on day 1, day 3 and day 6, in order to describe kinetics of evolution of soluble forms and ligands of RAGE levels. Undiluted pulmonary edema fluid samples will be collected in intubated patients only, and blood samples will be simultaneously gathered from indwelling arterial and central venous catheters. The concentrations of soluble forms (sRAGE, esRAGE) and ligands of RAGE (HMGB-1, S100A12, AGEs) will be measured in duplicate by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients under mechanical ventilation
* Patients within the first 24 hours after onset of ALI/ARDS according to the 1994 American-European Consensus Conference (AECC)

Exclusion Criteria:

* Pregnancy
* Acute exacerbation of diabetes
* Dialysis for end-stage kidney disease
* Alzheimer's disease
* Amyloidosis
* Evolutive neoplastic lesion

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Defined population
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Soluble forms (sRAGE, esRAGE) and ligands of RAGE (HMGB-1, S100A12, AGEs) levels in the plasma from ICU patients within the first 24 hours after onset of ALI/ARDS | within the first 24 hours after onset of ALI/ARDS

SECONDARY OUTCOMES:
To describe kinetics of evolution of soluble forms (sRAGE, esRAGE) and ligands of RAGE (HMGB-1, S100A12, AGEs) levels in ICU patients with or without ALI/ARDS: biomarkers levels in pulmonary edema fluid and plasma on day 1, day 3, and day 6 | on day 1, day 3, and day 6
To describe the plasma and pulmonary levels of soluble forms (sRAGE, esRAGE) and ligands of RAGE (HMGB-1, S100A12, AGEs) in the setting of ALI/ARDS. | on day 1, day 3, and day 6.
To test the correlation between soluble forms (sRAGE, esRAGE) and ligands of RAGE (HMGB-1, S100A12, AGEs) levels and net alveolar fluid clearance in patients within the first 24 hours after onset of ALI/ARDS. | within the first 24 hours after onset of ALI/ARDS
To decribe venous-to-arterial differences in soluble forms (sRAGE, esRAGE) and ligands of RAGE (HMGB-1, S100A12, AGEs) levels during ALI/ARDS. - | on day 1, day 3, and day 6.
To test the correlation between biomarkers levels (soluble forms (sRAGE, esRAGE) and ligands of RAGE (HMGB-1, S100A12, AGEs)) and CT-scan lung morphology in patients within the first 24 hours after onset of ALI/ARDS | within the first 24 hours after onset of ALI/ARDS
To describe soluble forms (sRAGE, esRAGE) and ligands of RAGE (HMGB-1, S100A12, AGEs) levels in ICU patients under mechanical ventilation (MV), in order to assess the influence of MV on these markers: biomarkers levels in pulmonary edema fluid and plasma | on day 1, day 3, and day 6
To test the prognostic value of soluble forms (sRAGE, esRAGE) and ligands of RAGE (HMGB-1, S100A12, AGEs) levels in ICU patients with ALI/ARDS: | on day 28
To test the correlation between biomarkers levels (soluble forms (sRAGE, esRAGE) and ligands of RAGE (HMGB-1, | on day 1, day 3, and day 6.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Jabaudon M, Blondonnet R, Roszyk L, Pereira B, Guerin R, Perbet S, Cayot S, Bouvier D, Blanchon L, Sapin V, Constantin JM. Soluble Forms and Ligands of the Receptor for Advanced Glycation End-Products in Patients with Acute Respiratory Distress Syndrome: An Observational Prospective Study. PLoS One. 2015 Aug 14;10(8):e0135857. doi: 10.1371/journal.pone.0135857. eCollection 2015. PMID 26274928